CLINICAL TRIAL: NCT06880822
Title: Effects of a Closed-Loop and Neuroplasticity-Based Mindfulness Program for Reducing Stress in Family Caregivers of People with Dementia: a Randomized Controlled Trial with a Process Evaluation
Brief Title: Closed-Loop and Neuroplasticity-Based Mindfulness Program for Family Caregivers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Patrick KOR Pui Kin, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSEARS20240722001
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Caregiving Stress
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Closed-Loop and Neuroplasticity-Based Mindfulness Program (Experimental)
  Interventions: Behavioral: Closed-Loop and Neuroplasticity-Based Mindfulness Program
- Traditional Mindfulness Program (Without the Closed-Loop Approach) (Active Comparator)
  Interventions: Behavioral: Traditional Mindfulness Program (Without the Closed-Loop Approach)
- Psychoeducation (Active Comparator)
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Closed-Loop and Neuroplasticity-Based Mindfulness Program — The intervention includes three weekly 90-minute face-to-face mindfulness training sessions and daily guided self-practice using a closed-loop, neuroplasticity-based mobile app over 8 weeks. Training integrates mindfulness practices (e.g., mindful eating, body scanning) to help caregivers apply mindfulness in daily life. During self-practice, participants listen to a lesson, monitor distractions, and refocus on their breathing. Initial trials start at 20 seconds, adjusting by 10% if focused or decreasing by 20% if distracted, helping participants regulate attention. Progress is stored to continue in later sessions, with instant feedback during trials and delayed feedback on overall progress. Facilitators provide weekly follow-ups via the app to monitor caregivers' progress.
  Arms: Closed-Loop and Neuroplasticity-Based Mindfulness Program
Behavioral: Traditional Mindfulness Program (Without the Closed-Loop Approach) — Family caregivers in the traditional mindfulness group will participate in general mindfulness practices (e.g., mindful eating, body scanning, and mindful walking) without the closed-loop approach. These practices aim to help caregivers learn mindfulness skills and integrate them into their everyday life. Sessions will be delivered through a mobile approach with the same group size, duration, and frequency as the intervention groups.
  Arms: Traditional Mindfulness Program (Without the Closed-Loop Approach)
Behavioral: Psychoeducation — Family caregivers in the control group will receive self-directed e-learning on dementia care with support from a registered nurse experienced in dementia care or elderly care. This group will serve as a control for socialization and interaction aspects with peers and the interventionist (nurse). The self-directed learning will be delivered through a mobile approach, maintaining the same group size, duration, and frequency as the intervention groups. Educational content will include brief sessions on dementia care, caregiving skills, and group sharing of caregiving tasks.
  Arms: Psychoeducation

SUMMARY:
The aim of this study is to evaluate the effectiveness of a closed-loop and neuroplasticity-based mindfulness program for reducing stress among family caregivers of people with dementia. Participants will be randomly assigned to one of three groups: the closed-loop and neuroplasticity-based mindfulness program, a traditional mindfulness program, or brief education on dementia care. The closed-loop and neuroplasticity-based mindfulness program will include three weekly face-to-face training sessions (90 minutes each) and daily guided self-practice over 8 weeks via a mobile application. The traditional mindfulness program will not include the closed-loop approach but will feature general mindfulness practices with the same group size, duration, and frequency as the closed-loop program. The family caregivers in the control group will receive self-directed e-learning on dementia care with support from a registered nurse experienced in dementia care or elderly care, maintaining the same group size, duration, and frequency as the intervention groups. Evaluations will be conducted at baseline (0 weeks), immediately post-intervention (8 weeks), and during a follow-up assessment (6 months). All groups will complete the same assessments at the same time points.

DETAILED DESCRIPTION:
Demanding caregiving tasks and uncertainty about disease progression cause high levels of stress in family caregivers of people with dementia (PWD), threatening their health and dyadic relationships. While mindfulness-based interventions (MBI) have shown promise in reducing stress, several limitations exist. Most studies used intensive training (weekly 150-minute sessions for 8 weeks), which was demanding for family caregivers and led to high attrition rates (10.5%-17.2%). Additionally, a wandering mind during practice has been the most challenging aspect of mindfulness. Traditional mindfulness practices lack quantifiable metrics of success or performance feedback, making engagement and long-term compliance difficult. Recent studies of online mindfulness programs found they typically duplicated real-world practices, encountering similar implementation challenges. Furthermore, the manualized protocol (e.g., 45 minutes of daily practice) was often unachievable for many caregivers, leading to frustration. Mindfulness training should adapt to individual abilities. To address these limitations, the investigators propose integrating a closed-loop and neuroplasticity-based approach in mindfulness training.

The study will recruit community-dwelling family caregivers of people with dementia from three local nongovernmental organizations (NGOs) providing dementia care services in Hong Kong. After eligibility assessment and consent, participants will be randomly assigned to one of three groups: the closed-loop and neuroplasticity-based mindfulness program, a traditional mindfulness program, or brief education on dementia care.

The closed-loop and neuroplasticity-based mindfulness program comprises three weekly face-to-face mindfulness training sessions (90 minutes each) and daily guided self-practice through a mobile application over 8 weeks. The face-to-face training will incorporate the mobile application and various mindfulness practices to help caregivers integrate mindfulness skills into daily life. Facilitators will provide weekly mobile device follow-up to monitor progress.

Family caregivers in the traditional mindfulness group will practice general mindfulness techniques without the closed-loop approach. These practices will be delivered through a mobile approach with identical group size, duration, and frequency as the intervention group.

The brief education on dementia care group will receive self-directed e-learning supported by an experienced registered nurse. This control group will maintain the same group size, duration, and frequency as the intervention groups. Educational content will include sessions on dementia care, caregiving skills, and group sharing.

Outcome measures include perceived caregiving stress (primary outcome), depressive symptoms, peace of mind, caregiving burden, dyadic relationship, dispositional mindfulness, physiological stress, neuropsychiatric symptoms, and caregiving-related productivity loss. Feasibility measures include eligibility and enrollment, attendance rate, self-practice engagement, and retention rate. Evaluations will occur at baseline (0 weeks), post-intervention (8 weeks), and follow-up (6 months). All groups will complete identical assessments at the same time points.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above;
* Family caregiver of an individual who has been living in the community with a confirmed medical diagnosis of any type of dementia (verified through NGO records or care recipient's medical records) for more than one year;
* Living in the same household as the care recipient;
* Providing care with daily contact of 4 hours or more.

Exclusion Criteria:

* Has participated in any structured mind-body intervention or structured psychosocial intervention within 6 months prior to recruitment;
* Has an acute psychiatric condition that is potentially life-threatening or would limit participation in the study (indicated by answering "yes" to any of the six questions on the Columbia Suicide Severity Rating Scale).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Perceived Caregiving Stress in the Family Caregiver | 6 months
  The Perceived Stress Scale (PSS) comprises 10 items rated on a 5-point Likert Scale (0 = never to 4 = very often) to assess perceived stress levels. The total score varies from 0 to 40, with a higher score reflecting more perceived stress. Scores within the ranges of 0-13, 14-26, and 27-40 correspond to low, moderate, and high levels of perceived stress, respectively.

SECONDARY OUTCOMES:
Depressive Symptoms in the Family Caregiver | 6 months
  The Center for Epidemiologic Studies Depression Scale (CESD) comprises 20 items rated on a 4-point Likert scale (0 = rarely or none of the time to 3 = most or almost all the time) to assess the severity of depressive symptoms experienced in the past week. The total score ranges from 0 to 60, with a higher score indicating more severe depressive symptoms. Scores within the ranges of 0-14, 15-21, and 22-60 correspond to low, mild to moderate, and a potential indication of major depression, respectively.
Peace of Mind in the Family Caregiver | 6 months
  The Peace of Mind Scale (PMS) consists of 7 items rated on a 5-point Likert scale (1 = not at all to 5 = all the time) that assess an internal state of peacefulness and harmony. Two items are reverse-scored. The total score ranges from 7 to 35, with higher scores indicating greater levels of peacefulness and harmony.
Caregiving Burden in the Family Caregiver | 6 months
  The Zarit Burden Interview (ZBI) consists of 22 items that measure the impact of caregiving on physical health, emotional well-being, social life, and financial status. Items are rated on a 5-point Likert scale (0 = never to 4 = nearly always). Total scores range from 0 to 88, with higher scores indicating greater caregiving burden.
Dyadic Relationship Between the Family Caregiver and the Care Recipient | 6 months
  The Dyadic Relationship Scale (DRS) measures the quality of the dyadic relationship between the family caregiver and the care recipient. This scale consists of two versions: the patient version (10 items) and the caregiver version (11 items). Both versions include two subscales: dyadic strain and positive dyadic interaction. They are rated on a 4-point Likert scale (1 = strongly disagree, 4 = strongly agree). Higher scores on each of these scales indicate higher levels of strain and positive interaction, respectively.
Dispositional Mindfulness in the Family Caregiver | 6 months
  The Mindful Attention Awareness Scale (MAAS) consists of 15 items that measure the core characteristics of dispositional mindfulness: receptive awareness and present-moment attention. Items are rated on a 6-point scale (1 = almost always to 6 = almost never). Total scores range from 15 to 90, with higher scores indicating greater levels of dispositional mindfulness.
Physiological Stress in the Family Caregiver | 6 months
  Physiological stress will be measured by heart rate variability (HRV) using the CorSense Heart Rate Variability Finger Sensor. HRV will be interpreted following the Guidelines for the Standard Measurement and Interpretation of HRV (European Society of Cardiology and the North American Society of Pacing and Electrophysiology) using the frequency-domain method.
Work Productivity and Activity Impairment in the Family Caregivers | 6 months
  The Work Productivity and Activity Impairment Questionnaire for Caregivers (WPAI:CG) consists of 6 items that measure productivity loss due to caregiving responsibilities. The questionnaire assesses four main outcomes: absenteeism (percentage of work time missed due to caregiving), presenteeism (percentage impairment while working due to caregiving), work productivity loss (percentage overall work impairment due to caregiving), and activity impairment (percentage activity impairment due to caregiving). The recall period is 7 days. Higher scores indicate greater impairment and less productivity. Total work productivity loss scores range from 0 to 100%, with higher percentages indicating greater impairment.
Neuropsychiatric Syndromes in the Care Recipient | 6 months
  The Neuropsychiatric Inventory (NPI) measures neuropsychiatric syndromes that occur in Alzheimer's disease and other neurodegenerative disorders. The NPI is administered by the family caregiver and consists of the following domains: Delusions, Hallucinations, Agitation/Aggression, Depression/Dysphoria, Anxiety, Elation/Euphoria, Apathy/Indifference, Disinhibition, Irritability/Lability, and Aberrant Motor Behavior. Each domain is rated based on its frequency (1 = rarely, less than once per week; 4 = very often, once or more per day) and severity (1 = mild, producing little distress in the patient; 3 = severe, very disturbing to the patient and difficult to redirect). A total score can be obtained for each domain by multiplying the frequency and severity ratings. The total score of the NPI is obtained by summing the scores across all domains, with a higher score indicating more severe neuropsychiatric syndromes.
Feasibility of Eligibility and Enrollment | 8 weeks
  Number of eligible participants, and the proportion of those eligible that enrolled will be assessed.
Feasibility of Attendance Rate | 8 weeks
  Number and proportion of attended participants.
Feasibility of Engagement to Self-Practice | 6 months
  Engagement with mindfulness practice will be determined by the duration of mindfulness practice as recorded through the participants' mobile application.
Feasibility of Retention Rate | 6 months
  Number and proportion of participants completing all assessments.

IPD SHARING:
Plan to Share IPD: Yes
The intervention protocol will be published.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Kor PPK, Chou KL, Tsang APL, Mak WWS, Galante J, Ho RTH, Wong SYS, Cheung DSK, Liu JYW, Zarit SH. Effects of a closed-loop mindfulness-based program for reducing stress in family caregivers of people with dementia: a study protocol of a randomized controlled trial. BMC Psychol. 2025 Jul 1;13(1):681. doi: 10.1186/s40359-025-02919-2. PMID 40597419